CLINICAL TRIAL: NCT02314637
Title: Long-term Safety Study of MP-513 as Monotherapy or in Combination With Sulfonylurea in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Long-term Safety Study of MP-513 as Monotherapy or in Combination With Sulfonylurea in Japanese Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-A8
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Results first posted 2015-01-02 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DPP-IV inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneligliptin (Experimental): Teneligliptin for 52 weeks
  Interventions: Drug: Teneligliptin
- Teneligliptin + Sulfonylurea (Experimental): Teneligliptin for 52 weeks in combination with sulfonylurea
  Interventions: Drug: Teneligliptin + Sulfonylurea

INTERVENTIONS:
Drug: Teneligliptin — Teneligliptin for 52 weeks
  Arms: Teneligliptin
Drug: Teneligliptin + Sulfonylurea — Teneligliptin for 52 weeks in combination with sulfonylurea
  Arms: Teneligliptin + Sulfonylurea

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MP-513 (Teneligliptin) as monotherapy or in combination with Sulfonylurea (glimepiride) in Japanese patients with type 2 Diabetes for 52 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

* In case of combination therapy with Sulfonylurea, patients who has been receiving a stable dose and regimen of sulfonylurea for diabetes over 12 weeks before administration of investigational drug
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* HbA1c criteria:

  * monotherapy: 6.9% - 10.5%
  * combination therapy with Sulfonylurea: 7.4 - 10.5%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients who are accepting treatments of arrhythmias
* Patients with serious diabetic complications
* Patients who are the excessive alcohol addicts
* Patients with severe hepatic disorder or severe renal disorder
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Reserch site, Shikoku, Japan

REFERENCES:
- [Result] Kadowaki T, Marubayashi F, Yokota S, Katoh M, Iijima H. Safety and efficacy of teneligliptin in Japanese patients with type 2 diabetes mellitus: a pooled analysis of two Phase III clinical studies. Expert Opin Pharmacother. 2015 May;16(7):971-81. doi: 10.1517/14656566.2015.1032249. Epub 2015 Apr 10. PMID 25861982

RESULTS

PARTICIPANT FLOW:
Groups:
- Teneligliptin + Sulfonylurea: Teneligliptin for 52 weeks in combination with sulfonylurea (glimepiride)
Period: Overall Study
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea
Started | 151 | 89
Completed | 135 | 75
Not Completed | 16 | 14
Not completed — Adverse Event | 4 | 8
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Other Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea | Total
Number analyzed (Participants) | 151 | 89 | 240
Age, Customized [Number; unit: participants]
  <65 years | 108 | 65 | 173
  >=65 years | 43 | 24 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 33 | 89
  Male | 95 | 56 | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) were defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after receiving the last dose of study drug.
Time Frame: 52 weeks
Population: Safety set, consisting of all patients, who received at least one dose of study drug and who had at least one safety data after the treatment of study drug.
Measure: Number; unit: participants
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea
Number analyzed (Participants) | 151 | 89
participants
  Serious Adverse Event | 6 | 7
  Other Adverse Event | 136 | 84

2. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Time Frame: Baseline and Week 52
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after the treatment of study drug. Analysis based on last observation carried forward, where the last postbaseline observed value was carried forward and used for Week 52 where data was missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea
Number analyzed (Participants) | 151 | 89
percent | -0.63 (0.67) | -0.81 (0.76)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 52
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea
Number analyzed (Participants) | 151 | 88
mg/dL | -12.4 (22.9) | -17.0 (30.5)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Teneligliptin | Teneligliptin + Sulfonylurea
Serious Adverse Events (participants affected / at risk) | 6/151 | 7/89
Other Adverse Events (participants affected / at risk) | 136/151 | 84/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin (N=151) | Teneligliptin + Sulfonylurea (N=89)
Diverticulitis (Infections and infestations) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin (N=151) | Teneligliptin + Sulfonylurea (N=89)
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 9 | 8
Cellulitis (Infections and infestations) | 1 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 3 | 2
Dermatitis infected (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Hordeolum (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 56 | 29
Onychomycosis (Infections and infestations) | 5 | 1
Otitis media (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 8 | 4
Pulpitis dental (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 7 | 2
Tonsillitis (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
Vulvovaginitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1
Myringitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 1 | 0
Cystitis bacterial (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 2 | 1
Latent syphilis (Infections and infestations) | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2
Thyroid mass (Endocrine disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 9
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 9
Schizophrenia (Psychiatric disorders) | 0 | 1
Somatoform disorder gastrointestinal (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 0
Migraine (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 2
Carotid arteriosclerosis (Nervous system disorders) | 3 | 0
Occipital neuralgia (Nervous system disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 4 | 0
Conjunctival granuloma (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 1
Diabetic retinopathy (Eye disorders) | 2 | 1
Dry eye (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1
Entropion (Eye disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Vertigo (Ear and labyrinth disorders) | 4 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 5 | 2
Dental caries (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 5 | 5
Gastritis (Gastrointestinal disorders) | 5 | 6
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Periodontal disease (Gastrointestinal disorders) | 2 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 1
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 8 | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Calculus prostatic (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Vaccination site dermatitis (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3
Albumin urine present (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 14 | 7
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 5 | 3
Blood triglycerides increased (Investigations) | 3 | 2
Blood uric acid increased (Investigations) | 4 | 2
Eosinophil count increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 5 | 3
Glucose urine present (Investigations) | 9 | 16
Blood urine present (Investigations) | 11 | 5
Monocyte count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 1
Protein urine present (Investigations) | 14 | 13
Urine ketone body present (Investigations) | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Occult blood positive (Investigations) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 3 | 1
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 3 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 9 | 5
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 2
Heat illness (Injury, poisoning and procedural complications) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other